CLINICAL TRIAL: NCT02334514
Title: The Effect of Oseltamivir Treatment on the Yield of Polymerase Chain Reaction Test for Confirmed Influenza Infection Among Adults - a Prospective, Cohort Study.
Brief Title: The Effect of Oseltamivir Treatment on the Yield of Polymerase Chain Reaction Test for Confirmed Influenza Infection
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, MICHAL PAUL md, M.D, Rambam Health Care Campus
Other Study IDs: 0472-14-RMB paul CTIL
Record Dates: First submitted 2015-01-01; First posted 2015-01-08 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Influenza
Keywords: Influenza; Viral shedding; oseltamivir; Polymerase Chain Reaction
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasopharyngeal swabs taken after start of oseltamivir treatment in patients diagnosed with influenza
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Adults with influenza: Patients diagnosed with influenza by PCR testing

SUMMARY:
The purpose of this study is to determine the duration of viral shedding in hospitalized patients with influenza virus, treated with oseltamivir.

DETAILED DESCRIPTION:
A prospective cohort study will be undertaken during the influenza season of 2015 in Rambam Medical Center, Haifa, Israel.

The study group will include inpatients older than 18 years, who have clinical presentation suggestive of influenza virus infection defined by the World Health Organization and the Center for Disease Control and Prevention, including sudden onset of high fever, cough, headache, muscle and joint pain, severe malaise, sore throat and runny nose, who were found positive to influenza virus by polymerase chain reaction test, and in whom anti viral treatment was indicated.

Exclusion criteria:

1. Immune compromised patients: patients after solid organ transplant, post bone marrow transplantation, with inherited or acquired immune deficiency, or patients treated chronically with immunosuppressive drugs.
2. Pregnant women.
3. Patients who were treated with oseltamivir in the previous 6 months.

Patients who approve their participation will to fill a questionnaire, and a polymerase chain reaction assay for influenza will be performed as follows:

The first sample will be taken right before the first dose of oseltamavir, and then on days 2, 3 and 5.

Samples will be stored at a temperature of +4 Celsius degrees for a maximum of 48 hours.

Outcomes: we will consider a positive polymerase chain reaction test 3 days after the initiation of treatment as prolonged shedding.

ELIGIBILITY:
Inclusion Criteria:

1. clinical presentation that suggest influenza virus infection, including sudden onset of high fever, cough, headache, muscle and joint pain, severe malaise, sore throat and runny nose,
2. positive to influenza virus by PCR test
3. anti viral treatment was indicated

Exclusion Criteria:

1. Immune compromised patients: patients after solid organ transplant, post bone marrow transplantation, with inherited or acquired immune deficiency, or patients treated chronically with immunosuppressive drugs.
2. Pregnant women.
3. Patients who were treated with oseltamivir in the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults hospitalized and diagnosed with influenza
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2014-11; Primary Completion 2017-05-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Duration of viral shedding in patients who were hospitalized with influenza infection. | 1 week
  PCR for influenza virus will be taken before the initiation of treatment, and at days 2, 3 and 5. Prolonged viral shedding will be defined as PCR positive at day 3.

CONTACTS AND LOCATIONS:
Overall Officials: Ami Neuberger, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel